CLINICAL TRIAL: NCT07154758
Title: Optimizing HF Treatment by Registry Screening for Need of Implementation and Referral to the Optimization Outpatient Clinic
Brief Title: Registry BAsed Optimization Of Therapy in Heart Failure
Acronym: REBOOT-HFrEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Gianluigi Savarese, MD, PhD, Region Stockholm
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-04364-01
Record Dates: First submitted 2025-08-15; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: Implementation; Guideline-directed medical therapy; registry; Swedish Heart Failure Registry
MeSH Terms: conditions — Heart Failure | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening through SwedeHF (Experimental): HFrEF patients enrolled in SwedeHF and screened for need of GDMT implementation through SwedeHF
  Interventions: Other: Screening for need of HFrEF GDMT implementation through SwedeHF
- Usual care (No Intervention): HFrEF patients not enrolled in the SwedeHF and therefore not undergoing screening for GDMT implementation

INTERVENTIONS:
Other: Screening for need of HFrEF GDMT implementation through SwedeHF — Screening for need of HFrEF GDMT implementation through SwedeHF
  Arms: Screening through SwedeHF

SUMMARY:
Rationale. Although several pharmacological treatments, namely renin-angiotensin-system inhibitors, sacubitril/valsartan, beta-blockers, mineralocorticoid receptor antagonists and sodium-glucose cotransporter-2 inhibitors, improve mortality/morbidity in heart failure with reduced ejection fraction (HFrEF), their use in clinical practice is still limited.

Aim. The aim of this project is to use the Swedish HF registry to identify HFrEF patients in need of 1) treatment implementation (initiation of treatments/uptitration), 2) screening and treatment of ID, and 3) with an indication for HF devices (CRT or ICD) but not implanted device, 4) referral for physiotherapy.

Outcomes.

Primary outcome: number of participants experiencing at least one of the following:

1. Drug initiation or uptitration (SGLT2i, MRA, BB, RASi, ARNi, iv iron)
2. ID screening
3. Referral for device therapy (CRT/ICD)

Secondary outcome:

1. Number of participants experiencing at least one drug initiation in the interventional vs. control arm.
2. Number of participants experiencing at least one drug dose up-titration in the interventional vs. control arm.
3. Number of participants experiencing referral for CRT or ICD in the interventional vs. control arm.
4. Number of participants screened for iron deficiency in the interventional vs. control arm.

Tertiary outcome:

1. Number of participants referred for physiotherapy in the interventional vs. control arm.

Study design. 500 patients will be screened through the Swedish Heart Failure Registry and, whether not on optimal medical treatment, implementation will be started. Outcome will be compared with a control population of 500 patients not enrolled in SwedeHF.

ELIGIBILITY:
Inclusion Criteria:

* Registration in SwedeHF with an index date after January 1st 2023 for the screening arm. For controls, hospital access after January 1st 2023.
* HF duration >6 months to ensure that patients had time to go through the treatment optimization process as recommended by the guidelines.
* HF with reduced EF (HFrEF) defined as categorical or continuous EF ≤40%
* Capable of giving signed informed consent (for the screening arm)

Exclusion Criteria:

* Under optimization of HF therapy
* In judgment of the investigator unlikely to understand or comply with study procedures

Control population is sex and age matched with the SwedeHF screening arm (1:1)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing at least one event of treatment optimization | End of implementation for the screening arm; 1-year from index date for the control arm
  Number of participants experiencing at least one of the following:
  1. Drug initiation or uptitration (SGLT2i, MRA, BB, RASi, ARNi, iv iron)
  2. ID screening
  3. Initiation/planning for device CRT/ICD Outcome measured as variable yes/no

SECONDARY OUTCOMES:
Number of participants experiencing at least one drug initiation in the interventional vs. control arm. | End of implementation for the screening arm; 1-year from index date for the control arm
  Number of participants experiencing at least one drug initiation (SGLT2i, MRA, RASi or ARNi, BB, iv iron) in the interventional vs. control arm.
Number of participants experiencing at least one drug dose up-titration in the interventional vs. control arm. | End of implementation for the screening arm; 1-year from index date for the control arm
  Number of participants experiencing at least one drug dose up-titration (MRA, RASi or ARNi, BB) in the interventional vs. control arm.
Number of participants experiencing referral for CRT or ICD in the interventional vs. control arm. | End of implementation for the screening arm; 1-year from index date for the control arm
  Number of patients referred for ICD/CRT in the interventional vs. control arm.
Number of participants screened for iron deficiency in the interventional vs. control arm. | End of implementation for the screening arm; 1-year from index date for the control arm
  Number of patients screened for ID in the interventional vs. control arm.

OTHER OUTCOMES:
Number of participants referred for physiotherapy in the interventional vs. control arm. | End of implementation for the screening arm; 1-year from index date for the control arm
  Referral for physiotherapy (Yes/No) in the interventional vs. control arm.

CONTACTS AND LOCATIONS:
Locations (6):
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hemse vårdcentral, Hemse
  - Länssjukhuset Ryhov, Jönköping
  - Karolinska University Hospital, Stockholm
  - St Görans hospital, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Swedish Heart Failure Registry webpage — https://www.ucr.uu.se/rikssvikt-en/